CLINICAL TRIAL: NCT07354061
Title: A Single-arm, Multicenter Clinical Study of Ensartinib Combined With Chemotherapy as Neoadjuvant Therapy for ALK-positive Non-small Cell Lung Cancer (NSCLC) (TD-ENSEMBLE Study)
Brief Title: Neoadjuvant Therapy With Ensartinib Combined With Chemotherapy for ALK-positive Non - Small Cell Lung Cancer (NSCLC)
Acronym: TD-ENSEMBLE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT202509-20-KYB-17-XWK
Record Dates: First submitted 2025-12-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
Keywords: Ensartinib; neoadjuvant; ALK - positive; Resectable
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ensartinib + Chemotherapy (Experimental)
  Interventions: Drug: Ensartinib + Chemotherapy

INTERVENTIONS:
Drug: Ensartinib + Chemotherapy — For patients with operable stage II - IIIB (N2) ALK - fusion - positive lung adenocarcinoma, after signing the informed consent form and being screened to meet the inclusion and exclusion criteria, they will receive treatment with ensartinib combined with pemetrexed and carboplatin for a duration of 9 weeks. Subsequently, after a comprehensive assessment, they will undergo surgical treatment. After the surgery, the pathological complete response rate (pCR), major pathological response rate (MPR), objective response rate (ORR), R0 resection rate, safety, etc. of the patients will be evaluated. Then, the researchers will decide whether the patients will receive post - operative adjuvant treatment according to the situation, until reaching the duration of post - operative adjuvant treatment, disease recurrence, death, loss to follow - up, or study termination, whichever occurs first.This study is divided into two stages. In Stage 1, 5 subjects will be enrolled as required to receive neo

SUMMARY:
The goal of this clinical trial is to learn if Ensartinib combined with chemotherapy works as a neoadjuvant treatment for patients with stage II-IIIB (N2) ALK-positive non-small cell lung cancer (NSCLC). It will also learn about the safety of this combination therapy. The main questions it aims to answer are:

* Does Ensartinib combined with chemotherapy lead to a pathological complete response (pCR) in surgically removed tumor tissue after neoadjuvant treatment?
* What medical problems do participants have when taking Ensartinib combined with chemotherapy? This is a single-arm study, meaning all participants will receive the investigational treatment. There is no placebo or active comparator group. The study will be conducted in two stages; the second stage will proceed only if no special, unexpected, or serious adverse events related to Ensartinib occur during the first stage involving 5 participants.

Participants will:

* Receive neoadjuvant treatment with Ensartinib (taken orally once daily) plus Pemetrexed and Carboplatin (administered intravenously every 3 weeks) for 9 weeks (3 cycles).
* Undergo surgical resection within 4 weeks after completing neoadjuvant therapy.
* Attend regular clinic visits for check-ups, blood tests, and imaging scans (CT, MRI) according to a detailed schedule during the neoadjuvant, surgical, and long-term follow-up periods (up to 10 years).
* Be monitored for adverse events and survival outcomes.

DETAILED DESCRIPTION:
The TD - ENSEMBLE Study: A Single - Arm, Multicenter Clinical Trial on Neoadjuvant Therapy with Ensartinib Combined with Chemotherapy for ALK - Positive NSCLC

Research Background

This is a clinical trial initiated by researchers. It aims to deeply analyze the current treatment landscape of non - small cell lung cancer (NSCLC), focusing on the unmet clinical needs of specific molecular subtype patient groups, and then conduct a study on the neoadjuvant therapy of ensartinib combined with chemotherapy for ALK - positive NSCLC.

Lung cancer is the leading cause of cancer - related deaths worldwide, and NSCLC accounts for approximately 80% of all lung cancer cases. For patients initially diagnosed with locally advanced (Stage II - III) NSCLC, surgical resection is a potentially curative treatment. However, even if the surgery is successful, the long - term survival rate of patients remains unsatisfactory. The 5 - year overall survival rate of patients with Stage II - IIIA NSCLC is about 36% to 60%. To improve the prognosis, platinum - based double - drug chemotherapy has become one of the standard treatment regimens for peri - operative (including neoadjuvant and adjuvant therapy) operable NSCLC. Large - scale meta - analyses have shown that compared with surgery alone, pre - operative neoadjuvant chemotherapy can increase the absolute 5 - year survival rate by about 5% and reduce the relative risk of death by 13%. However, the magnitude of this benefit is limited, indicating the need to explore more effective treatment strategies.

The study focuses on patients with NSCLC who have a positive anaplastic lymphoma kinase (ALK) fusion gene, which accounts for about 3% to 7% of all NSCLC cases. The development of ALK tyrosine kinase inhibitors (TKIs) has changed the treatment paradigm for advanced ALK - positive NSCLC. From the first - generation crizotinib to the subsequent second - and third - generation drugs, they have brought significant survival improvements for advanced patients. The study drug, ensartinib, is a second - generation ALK - TKI independently developed in China. It can not only strongly inhibit ALK but also has an inhibitory effect on the c - Met kinase. Clinical studies have shown that ensartinib has good efficacy in patients with advanced ALK - positive NSCLC who are resistant to crizotinib (the objective response rate (ORR) evaluated by independent review was 52%), and it has been approved for this indication. In the international multicenter Phase III eXalt3 study for first - line treatment, ensartinib significantly prolonged the median progression - free survival (mPFS was 31.3 months vs. 12.7 months) compared with crizotinib and has also been approved for first - line treatment.

Based on the excellent efficacy of ALK - TKIs in advanced diseases, applying them to the neoadjuvant treatment stage before surgery is a reasonable research direction. Some small - scale studies or case reports have explored the potential of ALK - TKIs for neoadjuvant treatment. For example, the SAKULA study (ceritinib), the NAUTIKA1 and ALNEO studies (alectinib), and the WILDERNESS study (brigatinib). These studies initially showed that ALK - TKI neoadjuvant treatment can achieve a relatively high major pathological response rate (MPR, about 42% - 66.7%) and pathological complete response rate (pCR, about 12% - 44.4%), and the safety is controllable. In addition, there are case reports of ensartinib achieving pCR in neoadjuvant treatment and retrospective analyses showing a trend of a high pCR rate of ensartinib combined with chemotherapy in neoadjuvant treatment.

Therefore, the TD - ENSEMBLE study aims to systematically evaluate the value of ensartinib (a targeted drug proven to be effective for advanced diseases) combined with a standardized chemotherapy regimen (pemetrexed + carboplatin) for the neoadjuvant treatment of operable early - stage (Stage II - IIIB, with N2 lymph node metastasis) ALK - positive lung adenocarcinoma patients.

Research Objectives and Evaluation Endpoints

* Primary Objective: To evaluate the pathological complete response rate (pCR) of the ensartinib - combined chemotherapy regimen. pCR is defined as the proportion of patients in whom no residual viable tumor cells are found in the resected primary tumor and metastatic lymph nodes after neoadjuvant treatment, as assessed by pathology. This is the gold standard for evaluating the depth of efficacy of neoadjuvant treatment.
* Secondary Objectives: To evaluate a series of other efficacy and safety indicators. The efficacy indicators include the major pathological response rate (MPR, the proportion of patients with residual viable tumor cells ≤10%), the objective response rate (ORR, evaluated by imaging according to the RECIST 1.1 criteria), the R0 resection rate (no cancer residue at the microscopic margin), the event - free survival (EFS, from enrollment to disease progression that hinders surgery, post - operative recurrence, metastasis, or death from any cause), the overall survival (OS, from enrollment to death from any cause), and the 3 - year EFS rate, 5 - year OS rate, and 10 - year OS rate. The safety objective is to evaluate the occurrence of adverse events of the combined regimen.
* Exploratory Objectives: To study potential biomarkers, including detecting the dynamic changes of minimal residual disease (MRD) before and after neoadjuvant treatment, analyzing the co - mutation status of other genes besides the ALK fusion at baseline, and analyzing the correlation between these factors and efficacy.

Study Design

* Study Type and Sample Size: A single - arm, multicenter, prospective, two - stage exploratory clinical study design is adopted. The planned total sample size is 20 patients, and the Simon's two - stage enrollment strategy is used. In the first stage, 5 patients are enrolled. After these 5 patients complete the neoadjuvant treatment and surgery, the safety data are reviewed by an independent data safety monitoring committee or the research team. If no special, unexpected, or serious adverse events (SAEs) related to ensartinib occur in these 5 patients during the neoadjuvant treatment, the study will proceed to the second stage, and the remaining 15 patients will be enrolled. If the above - mentioned safety problems occur, no new patients will be enrolled. The sample size calculation is based on the expected pCR rate of the primary endpoint. Referring to the previous pCR rate of approximately 4% in the general population with neoadjuvant chemotherapy, this study expects the ensartinib - combined chemotherapy to increase the pCR rate to 30%. Under the significance level (alpha = 0.025, one - sided) and test power (power = 90%), about 16 effective cases are required. Considering patient dropout, the final sample size is expanded to 20 to maintain sufficient statistical power.
* Study Process

  * Screening Period (within 28 days before enrollment): Potential subjects need to be strictly screened to confirm whether they meet the inclusion criteria and do not meet the exclusion criteria. Key screening steps include signing a written informed consent form; being histologically or cytologically diagnosed with lung adenocarcinoma through biopsy tissue (such as obtained by bronchoscopy or puncture); confirming the tumor to be ALK - fusion positive by methods recommended by the NCCN guidelines (such as PCR, FISH, IHC, or NGS); being confirmed as having operable Stage II - IIIB (N2) according to the AJCC 9th edition TNM staging system; having at least one measurable lesion that meets the RECIST 1.1 criteria confirmed by imaging (such as CT); having an ECOG performance status score of 0 or 1; undergoing comprehensive hematological, biochemical, and organ function tests to ensure the ability to tolerate treatment and surgery; evaluating cardiopulmonary function to confirm the feasibility of surgery; and conducting a pregnancy test for women of child - bearing potential. The protocol clearly defines detailed exclusion criteria, such as specific pathological types (squamous cell carcinoma, small cell carcinoma components), a history of previous anti - tumor treatment, active infections, severe or uncontrolled systemic diseases, a history of interstitial lung disease, specific cardiac criteria (such as QTc interval prolongation), pregnancy, or lactation.
  * Neoadjuvant Treatment Period (totaling 9 weeks): Enrolled patients receive a 9 - week neoadjuvant treatment. The treatment regimen is 225 mg of ensartinib taken orally once a day, combined with chemotherapy. Pemetrexed (500 mg/m²) and carboplatin (with the dose calculated according to the area under the blood - concentration - time curve (AUC) = 5 - 6) are administered intravenously on the first day of each 21 - day treatment cycle, for a total of 3 cycles. During this period, the safety and tolerability of patients are closely monitored. A blood routine test is performed once a week, and a blood biochemical test is performed once every 4 weeks (at the beginning of each cycle). At the end of the 9 - week treatment, patients undergo imaging evaluation (mainly enhanced chest CT) to assess the objective response of the tumor (ORR) according to the RECIST 1.1 criteria.
  * Surgical Period (within 4 weeks after the end of neoadjuvant treatment): A final imaging evaluation is performed 3 - 5 days after the completion of neoadjuvant treatment to determine the feasibility of surgery. After the evaluation, patients should undergo the planned surgical resection within 4 weeks, with the goal of achieving a complete R0 resection (no tumor cells at the microscopic margin). The resected tumor specimens are sent to the research center (such as the pathology department of the Second Affiliated Hospital of the Air Force Medical University, the leading unit, or the pathology departments of each sub - center) for standardized pathological processing and evaluation. Pathologists evaluate the proportion of residual viable tumor cells in the surgical specimens to determine the primary endpoint pCR and the secondary endpoint MPR. At the same time, surgical - related information, such as the surgical method and whether an R0 resection is achieved, is recorded.
  * Postoperative Follow - up Period

    * Safety Follow - up: A dedicated 30 - day safety follow - up is conducted for all patients after the last dose of the study drug to monitor new adverse events.
    * Survival Follow - up: After surgery, a long - term survival follow - up is entered to monitor disease recurrence and patient survival status. The follow - up plan is detailed. In the first year after surgery, outpatient re - examinations are carried out every 3 months; in the second and third years, every 4 months; in the fourth and fifth years, every 6 months; and once a year after 5 years. The re - examination contents include chest CT, abdominal CT, and serum tumor marker tests. Head MRI examinations are scheduled in the 6th and 12th months of the first year after surgery, the 4th month of the second year, and the 4th month of the third year. Bone scans are performed as clinically needed. The follow - up continues until disease recurrence/progression is confirmed, the patient withdraws informed consent, death occurs, the patient is lost to follow - up, or the study is terminated. Through this follow - up, long - term efficacy data such as event - free survival (EFS) and overall survival (OS) are collected.
* Efficacy Evaluation

  * Primary Efficacy Endpoint: The pathological complete response rate (pCR), that is, the proportion of patients in whom no viable tumor cells are found in the resected primary tumor and all regional lymph nodes after neoadjuvant treatment.
  * Secondary Efficacy Endpoints: Include the major pathological response rate (MPR, residual viable tumor cells ≤10%), the objective response rate (ORR, imaging - evaluated complete response (CR) + partial response (PR)), the R0 resection rate, the event - free survival (EFS), the overall survival (OS), and the survival rates at various time points (such as the 3 - year EFS rate and the 5 - year OS rate).
  * Safety Evaluation: All observed adverse events (AEs) and serious adverse events (SAEs) are graded for severity (grades 1 - 5) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI - CTCAE) Version 5.0. The causal relationship between AEs and the trial drug is judged by the investigator according to preset criteria (such as time sequence, known drug reaction types, de - challenge or re - challenge reactions), and is divided into five levels: "definitely related", "probably related", "possibly related", "possibly unrelated", and "unrelated". The protocol provides detailed definitions, reporting procedures, time limits (report within 24 hours), and handling principles for SAEs. It also provides the "Management Guidelines for Ensartinib Adverse Events", which gives specific dose adjustment and medical treatment suggestions for common adverse events.
* Data Analysis

  * Analysis Populations: Three analysis populations are defined. The full analysis set (FAS, the intention - to - treat (ITT) analysis set, including all subjects who signed the informed consent form and received at least one dose of the study drug. It is the main population for efficacy analysis. For missing efficacy endpoint data due to reasons such as withdrawal, the "last observation carried forward (LOCF)" method is used for imputation). The per - protocol set (PPS, a subset of the FAS, including subjects who strictly followed the study protocol, had good compliance, no major protocol deviations, and completed key evaluations. It is used to support the analysis results of the FAS and reflect the efficacy of the intervention under ideal conditions, serving as a sensitivity analysis). The safety analysis set (SAS, including all subjects who received at least one dose of the study drug and had at least one post - drug safety record. All safety analyses are based on this population).
  * Statistical Analysis Methods: Descriptive statistics are mainly used. For continuous variables (such as age, weight, and laboratory test values), the number of cases, mean, standard deviation, median, minimum, and maximum are used for description. For categorical variables (such as gender, ECOG score, tumor stage, and response status), frequency and percentage (composition ratio) are used for description. For the primary endpoint pCR rate and the MPR rate, ORR, and R0 resection rate in the secondary endpoints, the point estimate (the incidence in the sample) and its corresponding 95% confidence interval (CI) are calculated. For time - to - event endpoints (event - free survival EFS and overall survival OS), the Kaplan - Meier method is used for survival analysis. The median EFS and median OS (if the data are mature) are reported, and the survival rates at specific time points (such as the 3 - year EFS rate and the 5 - year OS rate) and their 95% CIs are calculated. For the safety analysis, all AEs and SAEs collected in the safety analysis set (SAS) are systematically summarized and listed. The incidence of AEs, the causal relationship with the study drug (the "definitely related", "probably related", and "possibly related" are combined and calculated as drug - related adverse reactions), the proportion of events leading to dose adjustment, suspension, or permanent discontinuation, and the outcome of events are reported by category (by organ system) and grade (by CTCAE 1 - 5).

Research Significance

The TD - ENSEMBLE study protocol is detailed and the design is rigorous, systematically planning each link from the project background to data statistical analysis. Through this single - arm, multicenter, prospective exploratory study, it aims to provide preliminary but crucial high - level evidence - based medical evidence for the efficacy (especially the pCR rate) and safety of ensartinib combined with chemotherapy for the neoadjuvant treatment of Stage II - IIIB (N2) ALK - positive non - small cell lung cancer, laying the foundation for subsequent possible confirmatory studies.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent prior to any study-specific procedures.
2. Aged between 18 and 75 years old (inclusive).
3. Histologically or cytologically confirmed lung adenocarcinoma via biopsy performed within 60 days prior to study enrollment.
4. Surgically resectable Stage II-IIIB (N2) lung adenocarcinoma (AJCC 8th Edition TNM Staging).
5. Confirmed ALK fusion mutation by detection methods recommended by NCCN guidelines.
6. Presence of at least one accurately measurable lesion, with the longest diameter ≥10 mm on baseline computed tomography (CT) scan (or lymph nodes with a short axis ≥15 mm) and suitable for accurate repeated measurements.
7. ECOG performance status of 0-1.
8. Adequate hematological, biochemical, and organ function:

   1. Hemoglobin ≥90 g/L (can be maintained or exceeded via transfusion);
   2. Absolute neutrophil count ≥1.5×10⁹/L;
   3. Platelet count ≥90×10⁹/L;
   4. Total bilirubin ≤2× upper limit of normal (ULN);
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× ULN;
   6. Creatinine ≤1.5× ULN; and creatinine clearance ≥60 mL/min.
9. Adequate cardiopulmonary function suitable for surgical treatment (assessed by ECG, echocardiography, pulmonary function tests, or blood gas analysis).
10. For female subjects of childbearing potential: Must use highly effective contraception for at least 2 weeks prior to initiation of study drug, have a negative pregnancy test, and not be breastfeeding at the start of dosing. Alternatively, must meet one of the following criteria at screening to demonstrate non-childbearing potential:

    1. Postmenopausal, defined as over 50 years old with amenorrhea for at least 12 months following cessation of all exogenous hormonal therapy.
    2. Women under 50 years old may be considered postmenopausal if they have amenorrhea for 12 months or more following cessation of exogenous hormone therapy and have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels within the postmenopausal range.
    3. Documented irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not including tubal ligation.
11. For male subjects with partners of childbearing potential: Must agree to use effective contraceptive methods during the study period and for 3 months after the last dose of study drug

Exclusion Criteria:

1. Presence of squamous cell carcinoma, large cell neuroendocrine carcinoma, or small cell carcinoma components.
2. Prior exposure to other anti-tumor therapies before enrollment.
3. Patient is pregnant or breastfeeding.
4. Current use of (or inability to discontinue use at least 3 weeks prior to receiving the first dose of study treatment) drugs or herbal supplements known to be strong inducers of CYP3A4. All patients must try to avoid concomitant use or ingestion of any drugs, herbal supplements, and/or foods known to have CYP3A4 induction effects.
5. Evidence of any severe or uncontrolled systemic disease, including uncontrolled hypertension and active bleeding, which in the investigator's opinion would compromise the patient's participation in the study or protocol compliance, or active infections including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
6. Prior history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any current evidence of active ILD.
7. History of hypersensitivity to active or inactive excipients of Ensartinib or drugs with similar chemical structures or classes to Ensartinib, as well as uncontrollable nausea and vomiting, chronic gastrointestinal diseases, inability to swallow formulated medication, or prior extensive bowel resection that would preclude adequate absorption of Ensartinib.
8. Intolerance to chemotherapy or refusal of chemotherapy.
9. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc) > 470 msec obtained from three ECGs using the screening ECG machine's QTc value.
   2. Any clinically significant abnormalities in rhythm, conduction, or morphology of resting ECG, such as left bundle branch block, third-degree heart block, or second-degree heart block.
   3. Any factors that increase the risk of QTc prolongation or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, unexplained sudden death under 40 years of age in first-degree relatives, or any concomitant medication known to prolong the QT interval.
10. History of definite neurological or psychiatric disorders, including epilepsy or dementia.
11. Any other conditions deemed by the investigator as unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | From enrollment to the end of treatment at 9 weeks

SECONDARY OUTCOMES:
Major pathological response rate (MPR) | From enrollment to the end of treatment at 9 weeks
Objective Response Rate (ORR) | From enrollment to the end of treatment at 3 years
R0 Resection Rate | Evaluated immediately after surgical intervention
3-year EFS Rate | Measured over a period of 3 years from study entry or treatment initiation
Event-Free Survival (EFS) | From enrollment to the end of treatment at 5 years
5-year OS Rate | Measured over a period of 5 years from study entry or treatment initiation.
Overall Survival (OS) | From enrollment to the end of treatment at 5 years
10-year OS Rate | Measured over a period of 10 years from study entry or treatment initiation.
Adverse events | from date of enrollment until the end of the study, assessed up to 60 months

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol